CLINICAL TRIAL: NCT06824597
Title: Impact of Baby Friendly Hospital Initiative Training Program on Nurses' and Mothers' Breastfeeding Practices and Experiences
Brief Title: Impact of Baby-friedly Hospital Initiative (BFHI) Training Program on Breastfeeding Practices
Acronym: BFHI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abeer Salah Ali Mohamed, Assistant Lecturer, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: breastfeeding
Record Dates: First submitted 2025-01-31; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Breastfeeding Outcomes
Keywords: training program - breastfeeding- practices-experiences

STUDY DESIGN:
Intervention Model Description: A quasi-experimental research design will be utilized. A quasi-experimental design is often described as a non-randomized, pre-post-intervention study, in which patients self-select into different treatments instead of being randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- training program for nurses (Experimental): The Baby Friendly Hospital Initiative training program will be conducted for maternity nurses at the inpatient postpartum wards (9, 10, 15 and 18) and the delivery unit in Mansoura University Hospital (MCH), Dakahlia governorate, Egypt.
  Interventions: Behavioral: Baby-friendly hospital initiative training program
- evaluating the outcome of the training program on breastfeeding mothers' practices (No Intervention): Before the training program, the first group of mothers (47 mothers) will be interviewed at the postpartum wards after delivery and the researcher will evaluate their self-reported breastfeeding practices during their hospital stay.
  After the training program, the second group (homogeneous) of mothers (47 mothers) will be interviewed at the postpartum wards after delivery and the researcher will evaluate their self-reported breastfeeding practices during their hospital stay.

INTERVENTIONS:
Behavioral: Baby-friendly hospital initiative training program — The Baby-Friendly Hospital Training Program is a critical intervention to improve maternal and infant health outcomes by promoting and supporting breastfeeding worldwide. It empowers the maternity nurses in this study to create an environment that prioritizes the needs of mothers and babies, ensuring the best possible start to life. It will be conducted for eight sessions (theoretical and practical), each session for about 20-30 minutes. It will include the importance of early initiation of breastfeeding, skin-to-skin contact immediately after birth, the importance of exclusive and continued breastfeeding, positions of breastfeeding, the importance of avoiding pre-lacteal feeds and unnecessary supplementation, advantages of rooming-in, and how to manage common breast and nipple conditions.
  The researcher will design an Arabic booklet and distribute it to the nurses at the first session as a guide to reinforce the teaching
  Arms: training program for nurses

SUMMARY:
This study aims to evaluate the impact of Baby Friendly Hospital Initiative training program on nurses' and mothers' breastfeeding practices and experiences.

Research Hypotheses

* Maternity nurses who participate in the Baby Friendly Hospital Initiative training program exhibit improvement in breastfeeding practice scores and more positive breastfeeding experiences after the training program than before.
* Breastfeeding mothers who receive Baby Friendly Hospital Initiative support have good breastfeeding practices and more positive breastfeeding experiences.

DETAILED DESCRIPTION:
Breastfeeding is a long-time investment in women's and babies' lives, not just a personal decision. World Health Organization (WHO) recommends breast milk as the most appropriate food for infants under six months of age. Breast milk contains all the nutrients that babies need in the first six months of life, so it is an ideal food for infants . Children who were breastfed had a lower risk of obesity and chest problems. Furthermore, breastfeeding mothers also benefited from breastfeeding, with lower rates of breast cancer, ovarian cancer, type II diabetes, and postnatal depression.

Exclusive breastfeeding (EBF) has been identified as the single most effective intervention for child survival, with the potential to prevent 13% of under-five deaths annually in low- and middle-income settings . WHO and United Nations Children's Fund (UNICEF) recommend optimal infant and young child feeding as immediate and early initiation of breastfeeding within the first hour of birth, EBF for the first 6 months of life, and with complementary feeding up to 2 years of age.

Early cessation of breastfeeding is a public health concern, especially in high-income countries, where only 25% of children were breastfeeding at 12 months of age, far below the global average of 74%. Women often cited difficulties, including low milk supply, painful nipples, and latching problems, as reasons for breastfeeding cessation. In addition, other factors, including lack of support or feeding advice, formula use, and returning to work, also contributed to breastfeeding cessation.

Evidence-based breastfeeding support is important for achieving breastfeeding recommendations, preventing morbidity and mortality, and promoting sustainable development goals. Thus, WHO and UNICEF have set a goal to increase breastfeeding rates to 75% in early infancy, 50% at six months, and 25% at one year of age.The Baby Friendly Hospital Initiative (BFHI) is a global program launched in 1991 by UNICEF and WHO to protect, promote and support breastfeeding in all maternity services. It requires all facilities that apply for the status of "Baby-Friendly Hospital" to provide maternity care to follow the "Ten Steps for the Successful Promotion of Breastfeeding" .

One of the 10 steps in this initiative is to have a written infant feeding policy that is routinely communicated to staff and parents. Step 2 requires the training of all healthcare staff in skills that are necessary to implement the policy. Healthcare providers play a key role in the beginning and continuity of the correct applications in breastfeeding and "Baby Friendly Hospital" criteria in society.In controlled studies, it was seen that training the nurses about BFHI principles increases their breastfeeding knowledge and practice scores and exclusive breastfeeding rates.

ELIGIBILITY:
Inclusion Criteria:

For nurses: all nurses who were working at inpatient postpartum wards and the delivery unit in Mansoura University Hospital with at least one year of work experience and who were providing direct care to the mothers and their newborns

For mothers:

* Who had the intention to breastfeed.
* Primiparous women
* Age between 18 and 35 years.
* Who had given birth to a singleton baby.
* Free from serious medical or obstetrical complications.

Exclusion Criteria:

* Breastfeeding mothers will be excluded from the study if their baby had:

  * Born before 37 weeks of gestation.
  * An Apgar score of less than 8 at 5 minutes.
  * A birthweight of less than 2,500 g.
  * Born with severe medical conditions or congenital malformations.
  * Admitted to the neonatal intensive care unit.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluating the nurses' experiences regarding baby-friendly hospital initiative training program | 3 months
  Interview questionnaire sheet will be adapted from (Gerhardsson, Oras, Mattsson, Blomqvist & Funkquist, 2022) and will be translated into Arabic by the researcher. It will consist of two parts: Part (1): Demographic and professional characteristics of the nurses. Part (2): Nurses' experiences regarding BFHI training program questionnaire: Before the training program, the nurses will be asked two questions: (Do you think breastfeeding is an interesting part of your job? / Do you think your role is important in improving breastfeeding support in the healthcare continuum). After the training program, the nurses will be asked whether their interest in breastfeeding increased during the training and whether they had received new tools that they could use when providing breastfeeding support.
Evaluating the nurses' practices regarding BFHI principles | 3 months
  Observational checklist to observe the nurses' practices regarding BFHI principles will be adapted from (Timalsina, 2020) and will consist of 10 items such as a demonstration of proper positioning, attachment, and rooming in….etc.
  Scoring system:
  The total practice score equals 10 and the nurses will be given a score (2) for done correctly, a score (1) for done incorrectly and a score (0) for not done. It will be classified into: poor for <50%, satisfactory 50-70%, and good practice >70%.

SECONDARY OUTCOMES:
Evaluating the secondary outcome of the training program for nurses on breastfeeding mothers' self- reported practices regarding the baby-friendly hospital initiative principles before and after the program. | 6 months
  Evaluating the impact of the training program on mothers' practices regarding the baby-friendly hospital initiative principles for one group of mothers before the training and another homogenous group after conducting the program and compare between the two groups. It will measure by:
  Structured Interview questionnaire will consist of two parts:
  Part (1): Demographic characteristics of the mothers Part (2): Self-reported BFHI practices questionnaire: This tool will be adapted from (WHO/UNICEF, 2009) to assess the self-reported breastfeeding practices that mothers experienced during the hospital stay such as time of initiation of breastfeeding, staff assistance with positioning and attaching the baby, expression of breast milk and skin to skin contact.
Evaluating the impact of the training program on mothers' experiences regarding breastfeeding | 6 months
  Evaluating the impact of the training program on mothers' experiences regarding breastfeeding for one group of mothers before the training and another homogenous group after conducting the program and compare between the two groups. It will measure by:
  Mothers' breastfeeding experiences questionnaire: This tool will be adapted from (Giannì et al., 2020). It will cover four areas: breastfeeding experience, breastfeeding difficulties, breastfeeding support, and intention to breastfeed again in the following pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Ali, Ass.lecturer, Principal Investigator — Faculty of Nursing, Mansoura University, Egypt
Locations (1):
- Faculty of Nursing, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Hawkins SS, Stern AD, Baum CF, Gillman MW. Compliance with the Baby-Friendly Hospital Initiative and impact on breastfeeding rates. Arch Dis Child Fetal Neonatal Ed. 2014 Mar;99(2):F138-43. doi: 10.1136/archdischild-2013-304842. Epub 2013 Nov 25. PMID 24277661
- [Background] Ducharme-Smith K, Gross SM, Resnik A, Rosenblum N, Dillaway C, Orta Aleman D, Augustyn M, Silbert-Flagg J, Caulfield LE. Exposure to Baby-Friendly Hospital Practices and Breastfeeding Outcomes of WIC Participants in Maryland. J Hum Lact. 2022 Feb;38(1):78-88. doi: 10.1177/0890334421993771. Epub 2021 Feb 16. PMID 33591853
- See also: Baby-friendly hospital initiative: revised, updated and expanded for integrated care. Section 4, Hospital self-appraisal and monitoring — https://apps.who.int/nutrition/publications/infantfeeding/bfhi_trainingcourse_s4/en/index.html